CLINICAL TRIAL: NCT04927780
Title: Perioperative Versus Adjuvant FOLFIRINOX for Resectable Pancreatic Cancer: the PREOPANC-3 Study
Brief Title: Perioperative or Adjuvant mFOLFIRINOX for Resectable Pancreatic Cancer
Acronym: PREOPANC-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Pancreatic Cancer Group (Unknown); Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Bas Groot Koerkamp, MD, PhD, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2021-0002; 2020-005141-16 (EudraCT Number)
Record Dates: First submitted 2021-06-08; First posted 2021-06-16 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Adenocarcinoma
Keywords: Neoadjuvant Therapy; Adjuvant Chemotherapy; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Pancreatic Neoplasms; Pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Leucovorin; Fluorouracil; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Perioperative mFOLFIRINOX (Experimental): Patients in the intervention arm (arm 1) start with neoadjuvant mFOLFIRINOX (consisting of oxaliplatin 85 mg/m², irinotecan 150 mg/m², leucovorin 400 mg/m², all at day 1, and fluorouracil continuous IV infusion 2.4 g/m² over 46 hours). Cycles are repeated every 14 days. After eight cycles, surgical resection is performed in the absence of unresectable or metastatic disease. After resection, four cycles of adjuvant mFOLFIRINOX are scheduled.
  Interventions: Drug: Leucovorin Calcium; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Oxaliplatin; Procedure: Resection
- Arm 2: Adjuvant mFOLFIRINOX (Active Comparator): Patients in the comparator arm (arm 2) start with surgery. After resection, 12 cycles of adjuvant mFOLFIRINOX (consisting of oxaliplatin 85 mg/m², irinotecan 150 mg/m², leucovorin 400 mg/m², all at day 1, and fluorouracil continuous IV infusion 2.4 g/m² over 46 hours) are scheduled.
  Interventions: Drug: Leucovorin Calcium; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Oxaliplatin; Procedure: Resection

INTERVENTIONS:
Drug: Leucovorin Calcium — IV
Drug: Fluorouracil — IV
Drug: Irinotecan Hydrochloride — IV
Drug: Oxaliplatin — IV
Procedure: Resection — Open or minimally-invasive pancreatectomy.

SUMMARY:
The PREOPANC-3 study is a randomized, multicenter, phase 3 trial. Patients with resectable pancreatic cancer will be randomly assigned (1:1) to 8 cycles of neoadjuvant mFOLFIRINOX followed by surgery and 4 cycles of adjuvant mFOLFIRINOX (arm 1) or to upfront surgery followed by 12 cycles of adjuvant mFOLFIRINOX (arm 2).

The primary objective of the trial is to determine whether perioperative mFOLFIRINOX improves overall survival compared with adjuvant mFOLFIRINOX in patients with resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically (Bethesda 5 or 6) confirmed pancreatic ductal adenocarcinoma.
* Resectable tumor according to Dutch Pancreatic Cancer Group criteria: no arterial contact and venous contact with the superior mesenteric vein or portal vein of 90 degrees or less
* No evidence for metastatic disease
* WHO performance status of 0 or 1
* Ability to undergo surgery and mFOLFIRINOX chemotherapy
* Leucocytes (WBC) ≥ 3.0 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin ≥ 6.0 mmol/l
* Renal function: eGFR ≥ 40 ml/min
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Prior radiotherapy, chemotherapy, or surgery for pancreatic cancer.
* Prior chemotherapy precluding mFOLFIRINOX.
* Previous malignancy (excluding non-melanoma skin cancer, pancreatic neuroendocrine tumor (pNET) <2cm, and gastrointestinal stromal tumor (GIST) <2cm), unless no evidence of disease and diagnosed more than 3 years before diagnosis of pancreatic cancer, or with a life expectancy of more than 5 years from date of inclusion.
* Pregnancy or lactation.
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years after randomization.
  The time between randomization and death from any cause. Patients alive at last follow-up are censored.

SECONDARY OUTCOMES:
Progression free survival | Up to 5 years after randomization.
  The time between randomization and locoregional progressive disease before or during treatment (resulting in irresectability), the occurrence of distant metastases, recurrent pancreatic cancer after surgery or death from any cause. Patients alive and free of these events at last follow-up are censored.
Distant metastases free survival | Up to 5 years after randomization.
  The time between randomization and the occurrence of distant metastases or death from any cause. Patients alive and free of these events at last follow-up are censored.
Locoregional progression free survival | Up to 5 years after randomization.
  The time between randomization and locoregional progression before or during treatment (resulting in irresectability), locoregional recurrence after resection or death from any cause. Patients alive and free of these events at last follow-up are censored.
Distant metastases free interval | Up to 5 years after randomization.
  The time between randomization and the occurrence of distant metastases. Distant metastases are considered an event and patients are censored at death or last follow-up when without this event.
Locoregional progression free interval | Up to 5 years after randomization.
  The time between randomization and locoregional progression before or during treatment (resulting in irresectability), or locoregional recurrence after resection. Locoregional progressive disease before or during treatment or locoregional recurrence after resection are considered an event and patients are censored at death or last follow-up when free of these events.
Chemotherapy start rate | 4 months
  The percentage of patients who received at least one cycle of scheduled chemotherapy.
Number of chemotherapy cycles received. | 9 months
  The number of mFOLFIRINOX cycles patients received.
Chemotherapy completion rate | 9 months
  The percentage of patients who completed all cycles of scheduled chemotherapy.
Dose intensity | 9 months
  The amount of drug delivered as a percentage of planned dose according to the protocol.
Staging laparoscopy rate | At the time of surgery.
  The percentage of patients that actually underwent a staging laparoscopy, regardless whether a surgical exploration or resection was performed.
Laparoscopy yield | At the time of surgery.
  The percentage of patients that underwent staging laparoscopy and were diagnosed with metastatic or unresectable disease during this procedure.
Surgical exploration rate | At the time of surgery.
  The percentage of patients who underwent a surgical exploration (open or minimally-invasive), regardless whether a resection was performed.
Resection rate | At the time of surgery.
  The percentage of patients that underwent a curative-intent resection.
Microscopically margin-negative (R0) resection rate | At the time of surgery.
  The percentage of patients that underwent a microscopically margin-negative (R0) resection. The resection is considered R0 if there is no tumor within 1 mm of the margins.
Lymph node-negative (N0) resection rate | At the time of surgery.
  The percentage of patients that underwent a resection with negative lymph nodes (N0) in the surgical specimen.
Pathologic response | At the time of surgery.
  Tumor regression score in the surgical specimen
Adverse events as assessed by the CTCAE version 5.0 | Until 30 days after last chemotherapy.
  Adverse events are assessed during neoadjuvant therapy and adjuvant therapy.
Postoperative complications | Up to 90 days after surgery.
  According to the Clavien-Dindo classification and by the International Study Group of Pancreatic Surgery and International Study Group of Liver Surgery.
Serum CA 19-9 and CEA response | 9 months
  The change in carbohydrate antigen 19-9 (CA 19-9) and carcinoembryonic antigen (CEA) after surgery and after 4, 8, and 12 cycles of mFOLFIRINOX compared to baseline.
Clinical response rate according to RECIST criteria version 1.1 | At the time of surgery.
  Response comparing baseline and restaging after 4 and 8 cycles of mFOLFIRINOX
Patient reported cancer-specific health-related Quality of Life (HRQoL) as assessed using the EORTC QLQ-C30 | Up to 5 years after randomization.
  At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year
Patient reported non-disease specific HRQoL as assessed using the EQ-5D-5L | Up to 5 years after randomization.
  At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year
Patient reported tumor-specific HRQoL as assessed using the EORTC LQPAN26 | Up to 5 years after randomization.
  At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year
Patient reported Quality of Life as assessed using the worry of progression of cancer scale (WOPS) | Up to 5 years after randomization.
  At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year
Patient reported chemotherapy-induced peripheral neuropathy as assessed using the EORTC QLQ-CIPN20 | Up to 5 years after randomization.
  At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year
Patient reported Quality of Life as assessed using the happiness, hospital, anxiety and depression scale (HADS) | Up to 5 years after randomization.
  At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year
Patient reported Quality of Life as assessed using Exocrine Pancreatic Insufficiency (EPI) questionnaire | Up to 5 years after randomization.
  At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year

CONTACTS AND LOCATIONS:
Overall Officials: Bas Groot Koerkamp, MD, PhD, Principal Investigator — Erasmus MC University Medical Center
Locations (22):
- Netherlands (18):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Meander Medical Center, Amersfoort
  - Amsterdam UMC, Amsterdam
  - OLVG, Amsterdam
  - Amphia Hospital, Breda
  - Deventer Hospital, Deventer
  - Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Tjongerschans Hospital, Heerenveen
  - Medical Center Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Maastricht UMC+, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC University Medical Center, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Regional Academic Center Utrecht, Antonius Hospital, Utrecht
  - Isala Hospital, Zwolle
- Oslo University Hospital, Oslo, Norway
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] van Dam JL, Verkolf EMM, Dekker EN, Bonsing BA, Bratlie SO, Brosens LAA, Busch OR, van Driel LMJW, van Eijck CHJ, Feshtali S, Ghorbani P, de Groot DJA, de Groot JWB, Haberkorn BCM, de Hingh IH, van der Holt B, Karsten TM, van der Kolk MB, Labori KJ, Liem MSL, Loosveld OJL, Molenaar IQ, Polee MB, van Santvoort HC, de Vos-Geelen J, Wumkes ML, van Tienhoven G, Homs MYV, Besselink MG, Wilmink JW, Groot Koerkamp B; Dutch Pancreatic Cancer Group. Perioperative or adjuvant mFOLFIRINOX for resectable pancreatic cancer (PREOPANC-3): study protocol for a multicenter randomized controlled trial. BMC Cancer. 2023 Aug 7;23(1):728. doi: 10.1186/s12885-023-11141-5. PMID 37550634